CLINICAL TRIAL: NCT04603521
Title: Retrospective Study of Patients Long-Term Survival of Obstructive Hypertrophic Cardiomyopathy (HCM)
Brief Title: Patients' Long-Term Survival of Obstructive Hypertrophic Cardiomyopathy (HCM)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000093; 000093-H
Record Dates: First submitted 2020-10-24; First posted 2020-10-27 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Cardiomyopathy; Obstructive Hypertrophic Cardiomyopathy
Keywords: HCM; Septal Myectomy; Surgical Intervention; Genetic Heart Disease; Natural History
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hypertrophic cardiomyopathy (HCM): Survival after Myectomy Operation

SUMMARY:
Background:

HCM is a genetic heart disease. It can cause fatigue, chest pain, or even death. For more than 50 years, a surgery called septal myectomy has been used to help people with this disease. Dr. Andrew G. Morrow originated the surgery and performed it more than 200 times at NIH starting in 1960. Researchers want to learn the long-term success of this surgery.

Objective:

To determine long-term survival at least 35 years after surgical myectomy at NIH and examine data for people who are confirmed to be deceased or alive.

Eligibility:

People who had surgical myectomy by Dr. Morrow from 1960 to 1983.

Design:

This study uses images and data that were obtained in the past. Many of the participants are deceased. Most of the others are no longer being followed at the NIH.

The medical records of people treated by Dr. Morrow were microfiched. These records can be accessed at the NIH. The records will be searched for keywords to find participants for this study.

Participants clinical data, such as lab testing and imaging, will be used. Other data collected as part of the original study will also be used.

Researchers will use participants name, date of birth, and Social Security number to learn if they are alive or deceased. If they are deceased, researchers will try to find the age of death. Online databases and search engines will also be used. Survival data will be compared to data from the general U.S. population for the same time period.

Data will be stored in a database that is password protected.

The study will last about 1 year.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a relatively common autosomal dominant genetic heart disease which may produce lifestyle limiting symptoms or even death. Medication can sometimes be of benefit, but surgical intervention with septal myectomy has been an alternative intervention. The experience with this surgery at NIH provides a unique opportunity to evaluate the long-term success of this operation.Dr. Andrew G. Morrow was the originator of this operation and performed over 200 septal myectomies at NIH starting in 1960. Reviewing the results of his experience will provide important information regarding the benefits of this intervention in these patients.

ELIGIBILITY:
* ELIGIBILITY:

Patients operated on 1960-1983 with surgical myectomy by Dr. Andrew G. Morrow at the NIH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients upon whom Dr. Andrew Morrow performed a surgical myectomy at the NIH between 1960 and 1983.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Long term survival after surgical myectomy at NIH | Enrolled NIH subjects 1960-1983
  To determine long-term survival at least 35 years after surgical myectomy at NIH. To examine survival data in those subjects in whom we can confirm a date of death or an indication that they are still alive.

SECONDARY OUTCOMES:
Cause of Death | End of Study
  To determine cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Rosing, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dorobantu L, Ticulescu R, Greavu M, Dermengiu A, Alexandrescu M, Trofin M. Current management and surgical advances in patients with hypertrophic obstructive cardiomyopathy. Kardiol Pol. 2019 Sep 23;77(9):829-836. doi: 10.33963/KP.14965. Epub 2019 Sep 9. PMID 31495825
- [Background] Maron BJ, Ommen SR, Semsarian C, Spirito P, Olivotto I, Maron MS. Hypertrophic cardiomyopathy: present and future, with translation into contemporary cardiovascular medicine. J Am Coll Cardiol. 2014 Jul 8;64(1):83-99. doi: 10.1016/j.jacc.2014.05.003. PMID 24998133
- [Background] Rastegar H, Boll G, Rowin EJ, Dolan N, Carroll C, Udelson JE, Wang W, Carpino P, Maron BJ, Maron MS, Chen FY. Results of surgical septal myectomy for obstructive hypertrophic cardiomyopathy: the Tufts experience. Ann Cardiothorac Surg. 2017 Jul;6(4):353-363. doi: 10.21037/acs.2017.07.07. PMID 28944176